CLINICAL TRIAL: NCT02300532
Title: Post-Marketing Surveillance of Gliadel 7.7mg Implant (All-case Observational Study)
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: GLI01S
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Malignant Glioma
Keywords: Malignant Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Patients with diagnosed malignant glioma treated by surgery, implanted Gliadel wafers 7.7mg
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Post-marketing surveillance to investigate the clinical safety and effectiveness in patients of all implantation of Gliadel with malignant glioma in the actual medical setting.

ELIGIBILITY:
Inclusion criteria:

* All-patient of Gliadel implantation

Exclusion criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed malignant glioma treated by surgery
Sampling Method: Non-Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2015-03-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events/Serious Adverse Events | Up to 3 months

SECONDARY OUTCOMES:
Survival rate | Up to 1 year
  Survival rate of subjects measured up to 1 year after implantation of Gliadel

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka, Osaka
  - Tokyo, Tokyo